CLINICAL TRIAL: NCT05459857
Title: A Randomised, Cross-Over, Nicotine Pharmacokinetic and Pharmacodynamic Study of Heated Tobacco Products Compared to Combustible Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NER01/0004
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product sequence ABCD (Experimental): Subjects use Product A on Day 1, Product B on Day 2, Product C on Day 3 and Product D on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence BDAC (Experimental): Subjects use Product B on Day 1, Product D on Day 2, Product A on Day 3 and Product C on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence CADB (Experimental): Subjects use Product C on Day 1, Product A on Day 2, Product D on Day 3 and Product B on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product sequence DCBA (Experimental): Subjects use Product D on Day 1, Product C on Day 2, Product B on Day 3 and Product A on Day 4
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D

INTERVENTIONS:
Other: Product A — Heated tobacco (HT) device with Intense HT sticks, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Other: Product B — Heated tobacco (HT) device with Regular HT sticks, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Other: Product C — Heated tobacco (HT) device with Menthol HT sticks, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Other: Product D — Subject's own brand combustible cigarette, used under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)

SUMMARY:
This is a randomised, cross-over, open-label, confinement study conducted in 24 adult male or female smokers of combustible cigarettes. The study investigates combustible and heated tobacco (HT) products in a cross-over design, including pharmacokinetic evaluation, subjective questionnaire assessments, as well as safety evaluation.

Subjects will perform a screening visit and a 5-day confinement period.

ELIGIBILITY:
Inclusion Criteria:

* Reports smoking an average of at least 10 manufactured combustible (menthol or non-menthol) cigarettes per day for at least 12 months prior to Screening
* Has a positive urine cotinine (>500 ng/mL) at Screening
* Has an exhaled carbon monoxide >10 ppm at Screening
* A female subject of childbearing potential must use contraception
* Male subject must use contraception

Exclusion Criteria:

* Has a history or presence of clinically significant disease or condition that, in the opinion of the Investigator, would jeopardise the safety of the subject or impact the validity of the study results.
* Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Screening
* Has a fever (>38.05°C) at Screening or check-in
* Has a history or presence of drug or alcohol abuse within 24 months of Check-in
* Pregnant or lactating females
* Has used any prescription smoking cessation treatments within 3 months prior to Check-in
* Is planning to quit smoking during the study or within the next 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Belfast, Nothern Ireland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Product Sequence ABCD | Product Sequence BDAC | Product Sequence CADB | Product Sequence DCBA
Started | 6 | 6 | 6 | 6
Completed | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Product Sequence ABCD | Product Sequence BDAC | Product Sequence CADB | Product Sequence DCBA | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.75) | 31.8 (8.11) | 49.2 (7.14) | 42.2 (12.5) | 41.0 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 2 | 10
  Male | 4 | 2 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Cmax
Description: Maximum measured plasma nicotine concentration, baseline-adjusted
Time Frame: 5 minutes pre-study product use and at 2, 4, 6, 8, 10, 15, 30, 45, 60, 120, and 240 minutes following the start of study product use
Population: The analysis population represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Product A: Subjects using Product A (Heated Tobacco device with Intense sticks), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product B: Subjects using Product B (Heated tobacco device with Regular sticks), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product C: Subjects using Product C (Heated tobacco device with menthol sticks), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product D: Subjects using Product D (subject's own brand combustible cigarette) for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 23 | 24 | 24 | 23
ng/mL | 10.500 (8.284) | 7.539 (4.653) | 8.191 (4.447) | 21.680 (10.810)

2. Primary Outcome: Nicotine AUCt
Description: The area under the concentration time curve for nicotine, from time 0 to the last observed non-zero concentration, baseline-adjusted
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 23 | 24 | 24 | 23
ng*min/mL | 746.00 (271.24) | 586.50 (192.03) | 585.00 (191.16) | 1514.00 (368.91)

3. Secondary Outcome: Urge to Smoke Pre-Use
Description: The subjects self-assess their urge to smoke by answering the question: "How strong is your current urge to smoke your usual brand cigarette?" on a Visual Analog Scale (VAS), with scores of 0 to 100, with 0 being 'not at all' and 100 being 'extreme'.
Time Frame: 10 minutes prior to the start of the product use session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 23 | 23 | 24 | 22
Units on a scale | 63.8 (27.4) | 57.8 (30.9) | 64.2 (29.6) | 62.8 (30.1)

4. Secondary Outcome: Urge to Smoke Post-Use
Description: as for outcome 3
Time Frame: At 240 min following the start of study product use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 24 | 24 | 24 | 23
units on a scale | 61.4 (28.4) | 67.5 (26.3) | 71.3 (21.7) | 67.5 (24.8)

5. Secondary Outcome: Smoking Urges Emax
Description: The subjects self-assess their urge to smoke at defined time points by answering the question: "How strong is your current urge to smoke your usual brand cigarette?" on a Visual Analog Scale (VAS), with scores of 0 to 100, with 0 being 'not at all' and 100 being 'extreme'. Emax is calculated as the maximum absolute value of change from baseline (i.e., the maximum response) in VAS scores.
Time Frame: 10 minutes prior to the start of the product use session, and at 4, 8, 15, 45, 60, 210 and 240 minutes following the start of study product use
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 23 | 23 | 24 | 22
units on a scale | 40.30 (25.75) | 32.90 (27.13) | 39.70 (29.72) | 49.80 (30.10)

ADVERSE EVENTS:
Time Frame: From screening until follow-up (7 days after the final product use)
Groups:
- Product A: Subjects using Product A (Heated Tobacco device Intense), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product B: Subjects using Product B (Heated tobacco device Regular), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
- Product C: Subjects using Product C (Heated tobacco device menthol), for one product use session, under controlled conditions (i.e., completely use a single unit of the product, with puffs taken at 30-second intervals and puffs 3 seconds in duration)
Arm/Group | Product A | Product B | Product C | Product D
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 2/24 | 3/24 | 1/24 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product A (N=24) | Product B (N=24) | Product C (N=24) | Product D (N=23)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 2 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT05459857/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT05459857/SAP_001.pdf